CLINICAL TRIAL: NCT03671148
Title: A Phase 3, Randomized, Double-Blind Study Comparing Risankizumab to Placebo in Subjects With Active Psoriatic Arthritis Including Those Who Have a History of Inadequate Response or Intolerance to Biologic Therapy(Ies) (KEEPsAKE 2)
Brief Title: A Study Comparing Risankizumab to Placebo in Participants With Active Psoriatic Arthritis Including Those Who Have a History of Inadequate Response or Intolerance to Biologic Therapy(Ies)
Acronym: KEEPsAKE2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M15-998; 2023-505477-33 (Other: EU CT)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Psoriatic Arthritis (PsA)
Keywords: KEEPsAKE 2; Risankizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab (Experimental): Participants randomized to receive 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1. At Week 24 participants will receive blinded placebo followed by open-label 150 mg risankizumab at Week 28, and every 12 weeks thereafter in Period 2 until the final dosing time point at Week 316.
  Interventions: Biological: Placebo; Biological: Risankizumab
- Placebo (Placebo Comparator): Participants randomized to receive double-blind placebo at Week 0, Week 4, and Week 16 in Period 1. At Week 24 participants will receive 150 mg risankizumab followed by open-label 150 mg risankizumab at Week 28, and every 12 weeks thereafter in Period 2 until the final dosing time point at Week 316.
  Interventions: Biological: Placebo; Biological: Risankizumab

INTERVENTIONS:
Biological: Placebo — Placebo for risankizumab administered by subcutaneous (SC) injection
Biological: Risankizumab — Risankizumab administered by subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of risankizumab in adults with moderately to severely active psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
The study consists of a Screening Period (approximately 35 days), Period 1, Period 2, and a 20-week Follow-up Period. Period 1 is a 24-week randomized, double-blind, placebo-controlled, parallel-group period. Period 2 is the long-term period and starts at Week 24. To maintain the blind to the original treatment allocation, treatment at the Week 24 Visit is blinded: participants randomized to placebo receive blinded risankizumab 150 mg, and participants randomized to risankizumab receive blinded placebo. At Week 28 and for the remaining dosing visits (to Week 316), all participants receive open-label risankizumab 150 mg every 12 weeks. Participants remain blinded to the original randomization allocation for the duration of the study. The total study duration is 336 weeks including a telephone call 140 days (20 weeks) after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriatic arthritis (PsA) with symptom onset at least 6 months prior to the Screening Visit and fulfillment of the Classification Criteria for PsA (CASPAR) at Screening Visit.
* Participant has active disease defined as ≥ 5 tender joints (based on 68 joint counts) and ≥ 5 swollen joints (based on 66 joint counts) at both the Screening Visit and Baseline.
* Diagnosis of active plaque psoriasis, with at least one psoriatic plaque of ≥ 2 cm diameter or nail changes consistent with psoriasis at Screening Visit.
* Participant has demonstrated an inadequate response or intolerance to biologic therapy(ies) or conventional synthetic disease modifying anti-rheumatic drugs (csDMARD) therapy(ies).

Exclusion Criteria:

* Participant is considered by investigator, for any reason, to be an unsuitable candidate for the study.
* Participant has a known hypersensitivity to risankizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (138):
- United States (55):
  - Pinnacle Research Group /ID# 167953, Anniston, Alabama
  - St. Jude Heritage /ID# 166842, Fullerton, California
  - Newport Huntington Medica /ID# 207423, Huntington Beach, California
  - Arthritis & Osteo Medical Ctr /ID# 166541, La Palma, California
  - East Bay Rheumatology Medical /ID# 166845, San Leandro, California
  - Inland Rheum Clin Trials Inc. /ID# 166621, Upland, California
  - Denver Arthritis Clinic /ID# 166442, Denver, Colorado
  - New England Research Associates, LLC /ID# 166525, Bridgeport, Connecticut
  - Yale University /ID# 166330, New Haven, Connecticut
  - Arthritis & Rheumatic Disease Specialties /ID# 212582, Aventura, Florida
  - SIMED Health, LLC /ID# 207457, Gainesville, Florida
  - Sweet Hope Research Specialty Inc /ID# 168163, Hialeah, Florida
  - Rheum Assoc of Central FL /ID# 201629, Orlando, Florida
  - HMD Research LLC /ID# 208428, Orlando, Florida
  - Millennium Research /ID# 201627, Ormond Beach, Florida
  - Arthritis Center, Inc. /ID# 208116, Palm Harbor, Florida
  - IRIS Research and Development, LLC /ID# 166351, Plantation, Florida
  - BayCare Medical Group /ID# 201630, St. Petersburg, Florida
  - West Broward Rheumatology Associates /ID# 201234, Tamarac, Florida
  - University of South Florida /ID# 208467, Tampa, Florida
  - ForCare Clinical Research /ID# 166375, Tampa, Florida
  - Arthritis and Rheumatology /ID# 169438, Atlanta, Georgia
  - Clinic of Robert Hozman/Clinical Investigation Specialists /ID# 166681, Skokie, Illinois
  - Springfield Clinic /ID# 166345, Springfield, Illinois
  - Ochsner Clinic Foundation /ID# 166622, Baton Rouge, Louisiana
  - The Arthritis & Diabetes Clinic, Inc. /ID# 166707, Monroe, Louisiana
  - MMP Women's Health /ID# 169334, Portland, Maine
  - Klein and Associates MD /ID# 166549, Hagerstown, Maryland
  - Duplicate_The Center for Rheumatology & Bone Research /ID# 166448, Wheaton, Maryland
  - Clinical Pharmacology Study Gr /ID# 166455, Worcester, Massachusetts
  - St. Paul Rheumatology /ID# 166599, Eagan, Minnesota
  - Clinvest Research LLC /ID# 166745, Springfield, Missouri
  - Clayton Medical Associates, P.C. dba Saint Louis Rheumatology /ID# 166389, St Louis, Missouri
  - Glacier View Research Institute /ID# 169344, Kalispell, Montana
  - Dartmouth-Hitchcock Medical Center /ID# 169443, Lebanon, New Hampshire
  - Ocean Rheumatology, PA /ID# 166561, Toms River, New Jersey
  - Arthritis Rheumatic and Back Disease Associates. P.A. /ID# 166658, Voorhees Township, New Jersey
  - Paramount Medical Research Con /ID# 166334, Middleburg Heights, Ohio
  - Health Research of Oklahoma /ID# 166408, Oklahoma City, Oklahoma
  - Altoona Ctr Clinical Res /ID# 166691, Duncansville, Pennsylvania
  - Clinical Research Ctr Reading /ID# 166354, Wyomissing, Pennsylvania
  - West Tennessee Research Institute /ID# 166429, Jackson, Tennessee
  - Nashville Arthritis and Rheumatology /ID# 208395, Nashville, Tennessee
  - Amarillo Ctr for Clin Research /ID# 208340, Amarillo, Texas
  - Tekton Research, Inc. /ID# 166493, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions /ID# 208156, Colleyville, Texas
  - Rheumatology Clinic of Houston /ID# 166636, Houston, Texas
  - West Texas Clinical Research /ID# 208155, Lubbock, Texas
  - SW Rheumatology Res. LLC /ID# 166587, Mesquite, Texas
  - Trinity Universal Research Associates, Inc /ID# 208387, Plano, Texas
  - DM Clinical Research /ID# 208350, Tomball, Texas
  - Kadlec Clinic Rheumatology /ID# 167667, Kennewick, Washington
  - Arthritis Northwest, PLLC /ID# 169535, Spokane, Washington
  - Rheumatology and Pulmonary Clinic /ID# 169341, Beckley, West Virginia
  - Rheumatic Disease Center, LLP /ID# 166682, Glendale, Wisconsin
- Argentina (7):
  - Hospital General de Agudos J. M. Ramos Mejia /ID# 169152, Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 208473, Ciudad Autonoma Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - DOM Centro de Reumatologia /ID# 208478, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Centro de Enfermedades del Hígado y Aparato Digestivo /ID# 169151, Rosario, Santa Fe Province
  - Instituto CAICI /ID# 169156, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia /ID# 208342, San Miguel de Tucumán, Tucumán Province
  - Cimer /Id# 169155, San Miguel de Tucumán
- Australia (5):
  - The Canberra Hospital /ID# 207591, Garran, Australian Capital Territory
  - Rheumatology Research Unit Sunshine Coast /ID# 207191, Maroochydore, Queensland
  - Griffith University /ID# 207504, Southport, Queensland
  - Emeritus Research /ID# 207195, Camberwell, Victoria
  - Monash Medical Centre /ID# 208033, Clayton, Victoria
- Belgium (4):
  - UZ Gent /ID# 210037, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 208209, Leuven, Vlaams-Brabant
  - ReumaClinic /ID# 208211, Genk
  - ZNA - Jan Palfijn /ID# 208210, Merksem
- Brazil (2):
  - CIP - Centro Internacional de Pesquisa /ID# 169524, Goiânia, Goiás
  - LMK Sevicos Medicos S/S /ID# 169541, Porto Alegre, Rio Grande do Sul
- Canada (5):
  - Percuro Clinical Research, Ltd /ID# 169530, Victoria, British Columbia
  - CIADS Research Co Ltd /ID# 169526, Winnipeg, Manitoba
  - Dermatrials Research /ID# 208303, Hamilton, Ontario
  - K. Papp Clinical Research /ID# 169527, Waterloo, Ontario
  - Centre Rhumatologie de l'Est /ID# 208302, Rimouski, Quebec
- Denmark (2):
  - Bispebjerg and Frederiksberg Hospital /ID# 168763, Frederiksberg, Capital Region
  - Aarhus University Hospital /ID# 168762, Aarhus C, Central Jutland
- Estonia (3):
  - East Tallinn Central Hospital /ID# 208317, Tallinn, Harju
  - MediTrials /ID# 207815, Tartu, Tartu
  - North Estonia Medical Centre /ID# 208319, Tallinn
- Finland (2):
  - Ite Pihlajanlinna Kuopio /ID# 208316, Kuopio
  - Turku University Hospital /ID# 208199, Turku
- France (2):
  - Duplicate_CHU Bordeaux-Hopital Pellegrin /ID# 211159, Bordeaux
  - CHRU Tours - Hopital Trousseau /ID# 209343, Chambray-lès-Tours
- Germany (4):
  - Rheumazentrum Ruhrgebiet /ID# 207212, Herne, North Rhine-Westphalia
  - Immanuel Krankenhaus Berlin /ID# 207214, Buch
  - Center of Innovative Diagnostics and Therapeutics (CIRI GmbH) /ID# 209494, Frankfurt
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH /ID# 209493, Hamburg
- Greece (3):
  - University General Hospital of Heraklion PA.G.N.I /ID# 206930, Heraklion, Crete
  - Naval Hospital of Athens /ID# 206928, Athens
  - Olympion General Clinic SA /ID# 207047, Pátrai
- Hungary (4):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 169248, Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 169237, Szeged, Csongrád megye
  - Vital-Medicina Kft. /ID# 208123, Veszprém, Veszprém megye
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 209054, Budapest
- Israel (5):
  - Sheba Medical Center /ID# 207468, Ramat Gan, Tel Aviv
  - Barzilai Medical Center /ID# 207471, Ashkelon
  - Rambam Health Care Campus /ID# 208169, Haifa
  - Meir Medical Center /ID# 207469, Kfar Saba
  - Rabin Medical Center /ID# 207470, Petah Tikva
- Italy (3):
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico di Modena /ID# 207800, Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 207268, Ancona
  - Azienda Ospedaliera Universitaria di Verona/Ospedale Borgo Roma /ID# 207264, Verona
- Netherlands (3):
  - Antonius Ziekenhuis /ID# 208581, Sneek, Provincie Friesland
  - Universitair Medisch Centrum Groningen /ID# 168450, Groningen
  - Medisch Centrum Leeuwarden /ID# 168449, Leeuwarden
- New Zealand (3):
  - Waikato Hospital /ID# 214276, Hamilton, Waikato Region
  - Middlemore Clinical Trials /ID# 214293, Auckland
  - CGM Research Trust /ID# 210596, Burwood Christchurch
- Poland (5):
  - Malopolskie Centrum Kliniczne /ID# 208011, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Reuma Park w Warszawie /ID# 210956, Warsaw, Masovian Voivodeship
  - Osteo-Medic S.C. /ID# 208013, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 208012, Gdansk, Pomeranian Voivodeship
  - Centrum Kliniczno-Badawcze /ID# 208014, Elblag, Warmian-Masurian Voivodeship
- Portugal (3):
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 208138, Ponte de Lima, Viana do Castelo District
  - Instituto Português De Reumatologia /ID# 208140, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 208139, Lisbon
- GCM Medical Group PSC - Hato Rey /ID# 208461, San Juan, Puerto Rico
- Changi General Hospital /ID# 208966, Singapore, Singapore
- South Africa (3):
  - Dr Jenny Potts /ID# 167628, Port Elizabeth, Eastern Cape
  - Arthritis Clinical Research Trials /ID# 167611, Cape Town, Western Cape
  - Winelands Medical Research Centre /ID# 167630, Stellenbosch, Western Cape
- Spain (5):
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 207822, Sabadell, Barcelona
  - Hospital Unversitario Marques de Valdecilla /ID# 208541, Santander, Cantabria
  - Hospital Universitario A Coruna - CHUAC /ID# 207819, A Coruña
  - Hospital Universitario 12 de Octubre /ID# 207820, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 207823, Valencia
- Sweden (4):
  - Duplicate_Karolinska Univ Sjukhuset /ID# 208174, Solna
  - Uppsala University Hospital /ID# 169098, Uppsala
  - Duplicate_Vastmanlands Sjukhus /ID# 168620, Västerås
  - Orebro Universitetssjukhuset /ID# 169400, Örebro, Örebro County
- United Kingdom (4):
  - Duplicate_Barts Health NHS Trust /ID# 210794, London, London, City of
  - Manchester University NHS Foundation Trust /ID# 207923, Manchester
  - Duplicate_Wirral University Teaching Hospital NHS Foundation Trust /ID# 210536, Metropolitan Borough of Wirral
  - Torbay and South Devon Nhs Foundation Trust /Id# 207926, Torquay

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Result] Ostor A, Van den Bosch F, Papp K, Asnal C, Blanco R, Aelion J, Alperovich G, Lu W, Wang Z, Soliman AM, Eldred A, Barcomb L, Kivitz A. Efficacy and safety of risankizumab for active psoriatic arthritis: 24-week results from the randomised, double-blind, phase 3 KEEPsAKE 2 trial. Ann Rheum Dis. 2022 Mar;81(3):351-358. doi: 10.1136/annrheumdis-2021-221048. Epub 2021 Nov 23. PMID 34815219
- [Derived] Gossec L, Balanescu A, D'Agostino MA, Ogdie A, Sewerin P, Deng Y, Shi L, Sugimoto Y, Zhong S, Xing Y, Lippe R, Kishimoto M. Efficacy of Risankizumab across distinct PsA phenotypes identified with machine learning analytics using data from biologic DMARD-Naive patients in two phase 3 clinical trials. Arthritis Res Ther. 2025 Nov 29;28(1):2. doi: 10.1186/s13075-025-03670-0. PMID 41318485
- [Derived] Ostor A, Van den Bosch F, Papp K, Keiserman M, Blanco R, Crowley A, White D, Biljan A, Madihlaba T, Carter K, Liu F, Soliman AM, Ashley D, Chen M, Glotfelty L, Kivitz A. Efficacy and Safety of Risankizumab for Active Psoriatic Arthritis: 196-Week Results from the KEEPsAKE 1 and KEEPsAKE 2 Randomized Clinical Trials. Rheumatol Ther. 2025 Dec;12(6):1103-1123. doi: 10.1007/s40744-025-00793-3. Epub 2025 Sep 30. PMID 41028616
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Risankizumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1403-1412. doi: 10.1007/s40744-024-00706-w. Epub 2024 Aug 9. PMID 39120849
- [Derived] Kwatra SG, Khattri S, Amin AZ, Ranza R, Kaplan B, Shi L, Padilla B, Soliman AM, McGonagle D. Enthesitis and Dactylitis Resolution with Risankizumab for Active Psoriatic Arthritis: Integrated Analysis of the Randomized KEEPsAKE 1 and 2 Trials. Dermatol Ther (Heidelb). 2024 Jun;14(6):1517-1530. doi: 10.1007/s13555-024-01174-4. Epub 2024 May 13. PMID 38739215
- [Derived] Ostor A, Van den Bosch F, Papp K, Asnal C, Blanco R, Aelion J, Carter K, Stakias V, Lippe R, Drogaris L, Soliman AM, Chen MM, Padilla B, Kivitz A. Efficacy and Safety of Risankizumab for Active Psoriatic Arthritis: 100-Week Results from the KEEPsAKE 2 Randomized Clinical Trial. Rheumatol Ther. 2024 Jun;11(3):633-648. doi: 10.1007/s40744-024-00657-2. Epub 2024 Mar 18. PMID 38498139
- [Derived] Ostor A, Van den Bosch F, Papp K, Asnal C, Blanco R, Aelion J, Lu W, Wang Z, Soliman AM, Eldred A, Padilla B, Kivitz A. Efficacy and safety of risankizumab for active psoriatic arthritis: 52-week results from the KEEPsAKE 2 study. Rheumatology (Oxford). 2023 Jun 1;62(6):2122-2129. doi: 10.1093/rheumatology/keac605. PMID 36282537
- [Derived] Thakre N, D'Cunha R, Goebel A, Liu W, Pang Y, Suleiman AA. Population Pharmacokinetics and Exposure-Response Analyses for Risankizumab in Patients with Active Psoriatic Arthritis. Rheumatol Ther. 2022 Dec;9(6):1587-1603. doi: 10.1007/s40744-022-00495-0. Epub 2022 Sep 30. PMID 36178584
- [Derived] Ostor AJK, Soliman AM, Papp KA, Padilla B, Wang Z, Eldred A, de Vlam K, Kivitz A. Improved patient-reported outcomes in patients with psoriatic arthritis treated with risankizumab: analysis of the Phase 3 trial KEEPsAKE 2. RMD Open. 2022 Jun;8(2):e002286. doi: 10.1136/rmdopen-2022-002286. PMID 35701011
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M15-998

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 99 sites in Argentina, Australia, Belgium, Brazil, Canada, Denmark, Estonia, France, Germany, Greece, Hungary, Israel, Italy, New Zealand, Poland, Portugal, South Africa, Spain, Sweden, United Kingdom, and the US including Puerto Rico.
  The study includes a 24-week double-blind placebo-controlled treatment period (Period 1) and an ongoing 184-week open-label treatment period (Period 2). Results are reported for Period 1 which was from 07 March 2019 to 22 June 2020.
Pre-assignment Details: Participants were randomized equally (1:1 ratio) to receive double-blind treatment with risankizumab 150 mg or matched placebo for 24 weeks. Randomization was stratified by current conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) use (0 vs ≥ 1), number of prior biologic therapies (0 vs ≥ 1), and extent of psoriasis (≥ 3% body surface area [BSA] or < 3% BSA) at Baseline.
Groups:
- Placebo: Participants randomized to receive placebo administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
- Risankizumab: Participants randomized to receive 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
Period: Overall Study
Arm/Group | Placebo | Risankizumab
Started | 220 | 224
Received Study Drug | 219 | 224
Completed (Completed Period 1 Study Participation) | 199 | 215
Not Completed | 21 | 9
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 7 | 2
Not completed — COVID-19 Logistical Restrictions | 0 | 1
Not completed — Other | 1 | 0
Not completed — Incomplete Randomization Visit | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
- Risankizumab: Participants received 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Risankizumab | Total
Number analyzed (Participants) | 219 | 224 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.64) | 53.1 (12.53) | 52.9 (12.57)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 176 | 178 | 354
  ≥ 65 years | 43 | 46 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 124 | 244
  Male | 99 | 100 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 42 | 85
  Not Hispanic or Latino | 176 | 182 | 358
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 210 | 218 | 428
  Black or African American | 3 | 2 | 5
  Asian | 3 | 2 | 5
  Multiple | 3 | 2 | 5
Current Use of Conventional Synthetic Disease-modifying Anti-rheumatic Drug (csDMARD) [Count of Participants; unit: Participants]
  Yes | 129 | 141 | 270
  No | 90 | 83 | 173
Number of Prior Biologic Therapies [Count of Participants; unit: Participants]
  0 prior biologics | 118 | 119 | 237
  ≥ 1 prior biologic | 101 | 105 | 206
Extent of Psoriasis [Count of Participants; unit: Participants] — The extent of psoriasis was measured by the physician as the total body surface area (BSA) involved with psoriasis. For purposes of clinical estimation, the total surface of the participant's palm and five digits was assumed to be approximately equivalent to 1% of BSA.
  Participants
    < 3% | 100 | 101 | 201
    ≥ 3% | 119 | 123 | 242
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness by pressure manipulation on physical examination.
  joints | 22.3 (13.80) | 22.8 (14.90) | 22.6 (14.35)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling by directed physical examination.
  joints | 13.6 (8.98) | 13.0 (8.73) | 13.3 (8.85)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to indicate the severity of their arthritis pain within the previous 24 hours using a horizontal 100 mm visual analog scale (VAS), ranging from 0 (no pain) to 100 (severe pain).
  score on a scale | 57.0 (23.09) | 55.0 (23.52) | 56.0 (23.30)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to rate their current psoriatic arthritis disease activity within the past 24 hours on a horizontal 100 mm VAS ranging from 0 (very well) to 100 (very poor).
  score on a scale | 56.2 (22.98) | 56.2 (21.79) | 56.2 (22.36)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: score on a scale] — The physician rated the participant's current global psoriatic arthritis disease activity in the past 24 hours (independently from the participant's assessment) on a 100 mm horizontal VAS ranging from 0 (very well) to 100 (very poorly). Population: participants with available data
  score on a scale
    number analyzed (Participants) | 213 | 219 | 432
    (all) | 60.7 (16.36) | 63.0 (17.01) | 61.9 (16.71)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: score on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week.
  Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  score on a scale | 1.13 (0.626) | 1.10 (0.618) | 1.12 (0.621)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 8.16 (17.120) | 7.45 (10.937) | 7.80 (14.319)
Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: score on a scale] — PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration, and desquamation of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked). The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). Population: Participants with psoriasis BSA involvement ≥ 3% at Baseline
  score on a scale
    number analyzed (Participants) | 119 | 123 | 242
    (all) | 8.35 (9.942) | 7.74 (6.698) | 8.04 (8.438)
Short-Form 36 (SF-36) Physical Component Summary (PCS) Score [Mean (Standard Deviation); unit: score on a scale] — The SF-36 Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS ranges from 0 to 100, with a normative mean value of 50; higher scores are associated with less disability.
  score on a scale | 35.16 (9.070) | 35.61 (8.766) | 35.39 (8.910)
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score [Mean (Standard Deviation); unit: score on a scale] — The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue, functional fatigue, emotional fatigue, and social consequences of fatigue. Participants respond to the questions on a scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue score is computed by summing the item scores, after reversing items worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue.
  score on a scale | 27.7 (12.71) | 28.2 (11.49) | 28.0 (12.10)
Presence of Enthesitis [Count of Participants; unit: Participants] — Enthesitis is inflammation of the entheses, the specific point where tendons or ligaments attach to bone. The Leeds enthesitis index (LEI) is a validated enthesitis index that uses 6 sites for evaluation of enthesitis: lateral epicondyle humerus left and right, Achilles tendon insertion left and right and medial condyle femur left and right. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 6 sites, for an overall score range of 0 to 6.
  Presence of enthesitis is defined as an LEI > 0.
  Participants
    Yes | 158 | 147 | 305
    No | 61 | 77 | 138
Presence of Dactylitis [Count of Participants; unit: Participants] — Dactylitis is characterized by swelling of the fingers or toes. The Leeds dactylitis index (LDI) basic is a score based on finger circumference and tenderness, assessed across all digits. The LDI basic measures the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference is multiplied by a tenderness score (1 for tender, 0 for non-tender). Scores for each digit are summed for the total LDI. The presence of dactylitis is defined as LDI > 0.
  Participants
    Yes | 57 | 40 | 97
    No | 160 | 184 | 344
    Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 24
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: Full analysis set; Non-responder imputation incorporating multiple imputation (MI) to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
percentage of participants | 26.5 [20.7 to 32.4] | 51.3 [44.8 to 57.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; The comparison between the risankizumab and placebo treatment groups for the primary efficacy endpoint (ACR20 at Week 24) was performed using the Cochran-Mantel-Haenszel (CMH) test adjusting for the stratification factors of current use of csDMARD (0 vs ≥ 1), number of prior biologic therapies (0 vs ≥ 1), and extent of psoriasis (≥ 3% BSA or < 3% BSA) at Baseline; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — A fixed sequence testing procedure is used to control the overall type I error rate at 2-sided alpha = 0.05 for the primary endpoint and ranked secondary endpoints; CMH test adjusted for the stratification factors of current use of csDMARD, number of prior biologic therapies, and extent of psoriasis at Baseline; Response Rate Difference = 24.5, 95% CI 2-sided [15.9 to 33.0] — Response Rate Difference = Risankizumab - Placebo

2. Secondary Outcome: Change From Baseline In Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 24
Description: The Health Assessment Questionnaire Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 24, excluding data after initiation of rescue medication or initiation of concomitant medications for psoriatic arthritis (PsA) use that could meaningfully impact efficacy assessment, was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
score on a scale | -0.05 [-0.12 to 0.02] | -0.22 [-0.28 to -0.15]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; MMRM analysis including treatment, visit, treatment-by-visit interaction, and stratification factors as fixed factors and Baseline value as covariate; Least Squares (LS) Mean Difference = -0.16, 95% CI 2-sided [-0.26 to -0.07] — Difference = Risankizumab - Placebo

3. Secondary Outcome: Percentage Of Participants Achieving Psoriasis Area Severity Index (PASI) 90 Response at Week 24
Description: PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration (thickening or hardening of the skin), and desquamation (peeling of the skin) of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked).
  The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline and Week 24
Population: Full analysis set participants with Baseline psoriasis BSA involvement ≥ 3%; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 119 | 123
percentage of participants | 10.2 [4.7 to 15.6] | 55.0 [46.2 to 63.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 44.3, 95% CI 2-sided [33.9 to 54.6] — Response Rate Difference = Risankizumab - Placebo

4. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: Full analysis set; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
percentage of participants | 25.3 [19.4 to 31.2] | 48.3 [41.7 to 54.8]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 22.6, 95% CI 2-sided [13.9 to 31.2] — Response Rate Difference = Risankizumab - Placebo

5. Secondary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) at Week 24
Description: A participant was classified as achieving MDA if 5 of the following 7 criteria were met:
  * Tender joint count (out of 68 joints) ≤ 1
  * Swollen joint count (out of 66 joints) ≤ 1
  * PASI score ≤ 1 (score ranges from 0 - 72) or percent BSA involved with psoriasis ≤ 3%
  * Patient's assessment of pain ≤ 15 (VAS from 0 to 100)
  * Patient's Global Assessment of disease activity ≤ 20 (VAS from 0 to 100)
  * HAQ-DI score ≤ 0.5 (index score ranges from 0 to 3)
  * Leeds Enthesitis Index ≤ 1 (assesses the presence or absence of enthesitis at 3 bilateral sites, for an overall score range from 0 to 6)
Time Frame: Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
percentage of participants | 11.4 [7.2 to 15.6] | 25.6 [19.9 to 31.4]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 14.0, 95% CI 2-sided [7.0 to 21.0] — Response Rate Difference = Risankizumab - Placebo

6. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The SF-36 PCS ranges from 0 to 100. A linear algorithm was applied to the calculation of the PCS which has a normative mean value of 50. Higher scores are associated with less disability; a score of 100 is equivalent to no disability and a score of 0 is equivalent to maximum disability. A positive change from Baseline score indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; a mixed effect model repeat measurement (MMRM) analysis with longitudinal data from observed cases up to Week 24, excluding data after initiation of rescue medication or initiation of concomitant medications for psoriatic arthritis use that could meaningfully impact efficacy assessment, was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
score on a scale | 2.01 [0.94 to 3.08] | 5.87 [4.86 to 6.88]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 3.86, 95% CI 2-sided [2.41 to 5.31] — Difference = Risankizumab - Placebo

7. Secondary Outcome: Change From Baseline In Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue (e.g., I feel tired), functional fatigue (e.g., trouble finishing things), emotional fatigue (e.g., frustration), and social consequences of fatigue (e.g., limits social activity). Participants respond to the questions on a scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
score on a scale | 2.6 [1.4 to 3.9] | 4.9 [3.7 to 6.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p = 0.009, Mixed Effect Model Repeated Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.2, 95% CI 2-sided [0.6 to 3.9] — Difference = Risankizumab - Placebo

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 24
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
percentage of participants | 9.3 [5.4 to 13.2] | 26.3 [20.3 to 32.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 16.6, 95% CI 2-sided [9.7 to 23.6] — Response Rate Difference = Risankizumab - Placebo

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 24
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 219 | 224
percentage of participants | 5.9 [2.7 to 9.0] | 12.0 [7.7 to 16.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p = 0.024, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 6.0, 95% CI 2-sided [0.8 to 11.3] — Response Rate Difference = Risankizumab - Placebo

10. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Week 24
Description: Resolution of enthesitis is defined as a Leeds Enthesitis Index (LEI) score = 0.
  LEI is an enthesitis measure developed specifically for PsA and assesses the presence or absence of tenderness at the following 3 bilateral enthesial sites: medial femoral condyles, lateral epicondyles of the humerus, and Achilles tendon insertions. Tenderness on examination is recorded as either present (coded as 1), absent (coded as 0), or not assessed for each of the 6 sites. The LEI is calculated by taking the sum of the scores from the 6 sites. The LEI ranges from 0 to 6 (worst).
Time Frame: Week 24
Population: Full analysis set participants with a Baseline LEI > 0; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 158 | 147
percentage of participants | 30.4 [23.2 to 37.6] | 42.9 [34.9 to 50.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 13.8, 95% CI 2-sided [3.5 to 24.2] — Response Rate Difference = Risankizumab - Placebo

11. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Week 24
Description: Resolution of dactylitis is defined as a Leeds Dactylitis Index (LDI) score = 0.
  The LDI basic is a score based on finger circumference and tenderness, assessed across all digits. The LDI basic measures the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference is multiplied by a tenderness score (1 for tender, 0 for non-tender). If both sides of a digit are considered involved, or the circumference of the contralateral digit cannot be obtained, a standard reference table is used.
  Scores from each digit are summed to provide the final LDI. A higher LDI indicates worse dactylitis.
Time Frame: Week 24
Population: Full analysis set participants with a Baseline LDI > 0; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 57 | 40
percentage of participants | 42.1 [29.3 to 54.9] | 72.5 [58.7 to 86.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 38.8, 95% CI 2-sided [22.9 to 54.8] — Response Rate Difference = Risankizumab - Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug to Week 24
Groups:
- Risankizumab 150 mg: Participants received 150 mg risankizumab administered by subcutaneous injection at Week 0, Week 4, and Week 16 in Period 1.
Arm/Group | Placebo | Risankizumab 150 mg
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/224
Serious Adverse Events (participants affected / at risk) | 12/219 | 9/224
Other Adverse Events (participants affected / at risk) | 11/219 | 17/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=219) | Risankizumab 150 mg (N=224)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=219) | Risankizumab 150 mg (N=224)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (13) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT03671148/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03671148/SAP_001.pdf